CLINICAL TRIAL: NCT03336138
Title: Application of Telemedicine to the Management of Aggressive Lymphomas: a Regional Comparative Study
Brief Title: Application of Telemedicine to the Management of Aggressive Lymphomas
Acronym: AMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/12/0072
Record Dates: First submitted 2017-10-30; First posted 2017-11-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMA group (Active Comparator): Patient with telephone follow-up modality called AMA (Assistance for ambulatory patients)
  Interventions: Other: AMA (Assistance for ambulatory patients)
- Control group (No Intervention): Patient with standard follow-up with no specific assistance for ambulatory patients

INTERVENTIONS:
Other: AMA (Assistance for ambulatory patients) — telephone follow-up modality
  Arms: AMA group

SUMMARY:
The purpose of this study is to evaluate the value of AMA in a comparative multicenter regional study as a reference for aggressive lymphoma. The primary endpoint will be RDI. This study consider that the AMA support should allow a significant improvement of the RDI compared to the control group and thus impact the duration without progression. The study covers 350 patients recruited from 10 regional centers.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a recent diffuse large B cell lymphoma (LBDGC), histologically proven, with treatment not started
* a priori likely to be treated by rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisolone every 21 days (R-CHOP21) for 8 cycles or rituximab, doxorubicin, cyclophosphamide, vindesine, bleomycin, and prednisone (R-ACVBP).
* Index international prognosis (IPI) measurable (IPI-aa), adjusted for age. Any IPI-aa is eligible.
* accepting the study

Exclusion Criteria:

* Patient with another type of lymphoma (including transformed follicular forms)
* Patient having already started his treatment.
* Life expectancy <3 months.
* Carcinologic history
* Serum positive for HIV or hepatitis B virus (HBV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
dose-relative intensity (RDI) | through study completion, an average of 2 years
  reduction of RDI

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT Guy, MD, Principal Investigator — University Hospital, Toulouse
Locations (10):
- France (10):
  - University Hospital of Toulouse, Toulouse, France
  - Clinique Claude Bernard, Albi
  - Hospital, Auch
  - Bayonne Hospital, Bayonne
  - University Hospital Bordeaux, Bordeaux
  - Hospital, Montauban
  - Clinique Marzet, Pau
  - Rodez Hospital, Rodez
  - Tarbes Hospital, Tarbes
  - Clinique Saint Jean, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lamy S, Bettiol C, Grosclaude P, Compaci G, Albertus G, Recher C, Nogaro JC, Despas F, Laurent G, Delpierre C. The care center influences the management of lymphoma patients in a universal health care system: an observational cohort study. BMC Health Serv Res. 2016 Aug 2;16(a):336. doi: 10.1186/s12913-016-1553-9. PMID 27485349
- [Result] Borel C, Lamy S, Compaci G, Recher C, Jeanneau P, Nogaro JC, Bauvin E, Despas F, Delpierre C, Laurent G. A longitudinal study of non-medical determinants of adherence to R-CHOP therapy for diffuse large B-cell lymphoma: implication for survival. BMC Cancer. 2015 Apr 15;15:288. doi: 10.1186/s12885-015-1287-9. PMID 25884669